CLINICAL TRIAL: NCT01354730
Title: A Pharmacovigilance Study for AdimFlu-S (A/H1N1) Influenza Vaccine in Pregnant Women
Status: Completed | Type: Observational
Sponsor: Adimmune Corporation (Industry)
Responsible Party: Daphne Shen, Adimmune Corporation
Other Study IDs: FLU10001
Record Dates: First submitted 2011-05-15; First posted 2011-05-17 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-05

CONDITIONS: Adverse Drug Reactions
Keywords: incidence; nature; seriousness; ADRs; vaccination
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Exposed cohort: The woman received AdimFlu-S (A/H1N1) vaccination between 2009/10 and 2010/02. The woman was pregnant at the time of vaccination.
- Unexposed cohort: The woman was gestation after April 2009.

SUMMARY:
This was a retrospective cohort study of pregnant women who had received the AdimFlu-S (A/H1N1) influenza vaccine during gestation period. Eligibility into the study was confirmed by chart review. If subject meets the eligibility criteria during the study period, data from the medical chart were extracted retrospectively from the date of vaccination and the infant (s) health status were followed until 8 weeks after the delivery.The unexposed cohort included pregnant women who did not receive any influenza vaccine during pregnancy. Within each participated study center, women who were gestation after April 2009 were randomly selected according to maternal age matching. The pregnancy outcome, including the status of delivery, abortion and gestational age, were extracted retrospectively by chart review.

ELIGIBILITY:
Inclusion Criteria:

Exposed Cohort:

* The woman received AdimFlu-S (A/H1N1) vaccination between 2009/10 and 2010/02.l
* The woman was pregnant at the time of vaccination.

Unexposed Cohort:

* The woman was gestation after April 2009.

Exclusion Criteria:

Exposed Cohort:

* Received any other H1N1 vaccination, e.g., Focetria.

Unexposed Cohort:

* The woman received any influenza vaccine during gestation period.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The target population was derived from medical centers in Taiwan: National Taiwan University Hospital, Chang Gung Memorial Hospital - LinKou and China Medical University Hospital.
  The sample size for this study was planned to include 500 cases in exposed cohort and 500 cases in unexposed cohort. Actual recruitment depended on the volume of pregnancy women received AdimFlu-S (A/H1N1) at each hospital. The size of unexposed cohort was be equal to the exposed cohort.
Sampling Method: Non-Probability Sample
Enrollment: 398 (Actual)
Dates: Start 2010-06; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The purpose of this study was to evaluate the incidence, nature and seriousness of adverse drug reactions (ADRs) occurring after vaccination. | 8 weeks after the delivery or abortion
  If subject meets the eligibility criteria during the study period, data from the medical chart were extracted retrospectively from the date of vaccination and the infant (s) health status were followed until 8 weeks after the delivery.